CLINICAL TRIAL: NCT06682728
Title: Adjuvant Sacituzumab Govitecan Plus Nivolumab in Patients with Muscle-Invasive Urothelial Carcinoma At High-Risk for Recurrence
Brief Title: Adjuvant Sacituzumab Govitecan and Nivolumab in Muscle-Invasive Urothelial Carcinoma At High-Risk Recurrence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Nataliya Mar, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4473; UCI 23-59 (Other: UCI CFCCC)
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma; Muscle-invasive Bladder Cancer
Keywords: UC; Urothelial Carcinoma; muscle-invasive urothelial carcinoma; MIBC; sacituzumab govitecan; nivolumab
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — sacituzumab govitecan; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sacituzumab Govitecan PLUS Nivolumab (Experimental): Patients eligible for this study treatment will receive combination therapy with Sacituzumab Govitecan with Nivolumab for 4 cycles, followed by single-agent Nivolumab for an additional 11 cycles.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Nivolumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Given IV
Drug: Nivolumab — Given IV

SUMMARY:
This is a phase 2 study, single-arm study of adjuvant combination therapy with Sacituzumab Govitecan and Nivolumab in patients with muscle-invasive urothelial carcinoma of the bladder, ureter, or upper tract, who are high risk for cancer recurrence post curative-intent surgery based on surgical pathology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of study consent.
* ECOG Performance Status of 0, 1 or 2 (see Appendix A).
* Histologically confirmed muscle-invasive UC originating in the bladder, ureter, or renal pelvis. Variant histology, except small cell carcinoma, is allowed.
* Underwent curative-intent surgery (i.e. RC or nephroureterectomy), performed within 180 days prior to study treatment initiation.
* Radiographic disease-free status as determined by imaging within 28 days of C1D1 of study treatment.
* Prior platinum-based NAC is allowed. If chemotherapy-naive, patient must be Cisplatin-ineligible (based on Galsky et al 2011 [10]) or refuse platinum AC.
* Prior treatment with neoadjuvant investigational agents is allowed (except PD-1/PD-L1 inhibitors or sacituzumab govitecan). No washout from neoadjuvant therapy is required.
* If NAC was given, patient must be considered at high risk for cancer recurrence due to having pathologic T2, T3, T4, or N+ disease on RC or nephroureterectomy surgical spec-imen.
* If no NAC was given, patient must be considered at high risk for cancer recurrence due to having pathologic T3, T4, or N+ disease on RC or nephroureterectomy surgical speci-men.
* Adequate organ and marrow function as defined below:
* ANC ≥ 1000/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 × institutional ULN (or ≤ 3.0 × ULN for subjects with Gilbert's disease)
* AST/ALT ≤ 3 × institutional ULN
* Alkaline phosphatase ≤ 3 × institutional ULN
* Serum albumin ≥ 2.8 g/dL
* Creatinine Creatinine clearance of ≥30 mL/min (calculated with Cockroft-Gault formula)
* Hemoglobin ≥ 9.0 g/dL
* aPTT ≤ 1.5 × institutional ULN
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (i.e. barrier methods including male condom, female condom, or diaphragm with spermicidal gel, etc.) that are approved by the Investigator. Contra-ception must be used during the course of the treatment and for 6 months after the last dose of study treatment.
* Female subjects of childbearing potential must not be pregnant following signing the study consent form. Female subjects are considered to be of childbearing potential unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal sta-tus (defined as at least 12 months of amenorrhea in a woman ≥ 45 years-of-age in the ab-sence of other biological or physiological causes).
* Recovery to ≤ Grade 1 of CTCAE version 5 toxicities related to any prior treatment for UC, unless the AE(s) is clinically non-significant and/or stable on supportive therapy as per discretion of the Investigator.
* Subjects with any type of genitourinary catheters (i.e. nephrostomy, Foley, etc) are al-lowed.
* Ability to understand and the willingness to sign a written informed consent. Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, hard of hearing, and illiterate individuals are eligible for this trial.

Exclusion Criteria

* Underwent a partial cystectomy or partial nephrectomy.
* History of adjuvant platinum-based chemotherapy or any other type of adjuvant therapy, including investigational agents, following surgical removal of UC.
* History of treatment with PD-1/PD-L1 inhibitors or sacituzumab govitecan prior to study treatment initiation.
* History of previous radiation therapy for treatment of UC.
* Radiographic evidence of metastasis.
* Receipt of or planning to receive any other concurrent investigational agents.
* History of active, known, or suspected autoimmune disease.
* Conditions requiring treatment with either systemic high-dose corticosteroids (e.g. prednisone dose of ≥ 10 mg or equivalent) or other immunosuppressive medications within 14 days of study treatment initiation.
* Inhaled or topical steroids are permitted in the absence of active autoimmune dis-ease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Major surgery within 28 days or minor surgery within 14 days before the first dose of study treatment. Subjects must have complete wound healing and resolution from complications of major or minor surgery before first dose of study treatment.
* Active malignancy within 3 years of study entry, except treated localized non-melanoma skin cancer, Gleason 6 prostate cancer on active surveillance, or curatively treated in situ cancer of the breast or cervix.
* Patients who do not have adequate organ and marrow function, as defined in Section 4.1 above.
* Uncontrolled intercurrent illness including, but not limited to, the following conditions:
* Active and/or uncontrolled bacterial, viral, or fungal infection within 7 days of study treatment initiation.
* History of HIV infection with detectable viral load.
* History of Hepatitis B or C infection with detectable viral load.
* History of severe liver impairment (Child-Pugh C liver cirrhosis).
* History of active tuberculosis (Bacillus tuberculosis).
* Congestive heart failure New York Heart Association (NYHA) Class 3 or 4, unstable angina pectoris, or serious uncontrolled cardiac arrhythmias.
* Stroke (including transient ischemic attack (TIA), myocardial infarction (MI), or other ischemic arterial event within 90 days before first dose of study treatment.
* Severe, uncontrolled bleeding within 14 days before first dose of study treatment.
* Uncontrolled diarrheal illness ≥ Grade 3 in severity within 14 days before first dose of study treatment.
* History of inflammatory bowel disease (i.e. ulcerative colitis, Crohn's disease, etc.) or any other condition that puts patients at high risk of developing severe diarrhea.
* Psychiatric illness/social situations causing inability to comply with study proce-dures or follow up.
* Pregnancy at the time of or following study consent.
* Breastfeeding at the time of or following study consent.
* Received a live vaccine within 28 days prior to the first dose of study treatment.
* Known or suspected severe hypersensitivity (Grade ≥ 3) to nivolumab, sacituzumab govitecan, irinotecan, and/or any of their components.
* History or current evidence of any condition, therapy, or laboratory/radiographic abnormal-ity that might confound the results of the study, interfere with the patient's ability to participate for the full duration of the study, or is not in the best interest of the patient to partici-pate in the study, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 6 months after last patient enrollment
  To determine investigator-assessed disease-free survival (DFS) at 6 months.

SECONDARY OUTCOMES:
Secondary (1) | Time from Cycle1 Day 1 of study treatment to first occurrence of a disease free survival event, up to 5 years.
  To determine investigator-assessed DFS (i.e. time from Cycle 1 Day 1 (C1D1) of study treatment to first occurrence of a DFS event), defined as any of the following:
  1. Local (pelvic) recurrence of UC (including regional lymph nodes)
  2. Urinary tract recurrence of UC (including all pathological stages and grades)
  3. Distant metastasis of UC
  4. Death from any cause
Secondary (2) | Time from Cycle 1 Day 1 of study treatment to diagnosis of distant metastases or death from any cause, up to 5 years.
  To determine investigator-assessed distant metastasis-free survival (MFS) (i.e. time from Cycle 1 Day 1 of study treatment to diagnosis of distant metastases or death from any cause).
Secondary (3) | Time from C1D1 of study treatment to death of any cause, up to 5 years.
  To determine overall survival (OS) (i.e. time from Cycle 1 Day 1 of study treatment to death of any cause).
Secondary (4) | Up to 5 years
  To determine incidence of Grade 3 or higher AEs.
Secondary (5) | Conversion from positive ctDNA to negative at any point from baseline assessment, up to 5 years.
  To determine rate of ctDNA clearance in ctDNA positive patients (i.e. conversion from positive ctDNA to negative at any point from baseline assessment).
Secondary (6) | Up to 5 years
  To perform exploratory biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Mar, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No